CLINICAL TRIAL: NCT01243073
Title: A Phase II Trial to Evaluate the Activity of Imetelstat (GRN163L) in Patients With Essential Thrombocythemia or Polycythemia Vera Who Require Cytoreduction and Have Failed or Are Intolerant to Previous Therapy, or Who Refuse Standard Therapy
Brief Title: Open Label Study to Evaluate the Activity of Imetelstat in Patients With Essential Thrombocythemia or Polycythemia Vera
Acronym: ET/PV
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Geron Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP14B015
Record Dates: First submitted 2010-11-11; First posted 2010-11-18 (Estimated); Last update posted 2016-01-26 (Estimated); Status verified 2015-12

CONDITIONS: Essential Thrombocythemia; Polycythemia Vera
Keywords: imetelstat; imetelstat sodium; GRN163L; telomerase inhibitor; telomerase; essential thrombocytosis; essential thrombocythemia; ET; polycythemia vera; PV
MeSH Terms: conditions — Thrombocythemia, Essential; Polycythemia Vera | interventions — imetelstat

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- imetelstat (Experimental): Induction dosing of 9.4 mg/kg weekly, followed by intermittent maintenance dosing.
  Interventions: Drug: Imetelstat

INTERVENTIONS:
Drug: Imetelstat

SUMMARY:
This is a phase II open-label study of single agent imetelstat in patients with essential thrombocytopenia or with polycythemia vera who have failed or are intolerant to at least one prior therapy, or who refuse standard therapy.

DETAILED DESCRIPTION:
For patients with ET: To obtain a preliminary estimate of efficacy of imetelstat, as measured by best hematologic response within the first year of therapy in patients with ET who have failed or are intolerant to at least one prior therapy, or who have refused standard therapy.

For patients with PV: To obtain a preliminary estimate of efficacy of imetelstat, as measured by maintenance of Hct < 45% in men and < 42% in women (or pre-specified Hct count that is tolerable) without phlebotomy or myelosuppressive therapy within the first year of therapy in patients with PV who have failed or are intolerant to at least one prior therapy, or who have refused standard therapy.

ELIGIBILITY:
Inclusion Criteria:

ET-Specific Criteria

* Confirmed diagnosis of ET by WHO criteria
* Patients with ET requiring cytoreduction who have failed or are intolerant to at least one prior therapy, or who refuse standard therapy
* Laboratory criteria (within 14 days of first study drug administration):

  * Platelets > 600,000/μL
  * ANC ≥ 1500/μL
  * Hemoglobin ≥ 10 g/dL

PV-Specific Criteria

* Confirmed diagnosis of PV by WHO criteria
* Patients with PV requiring cytoreduction with phlebotomy and/or myelosuppressive agents

  * Patients may have failed or are intolerant to at least one prior therapy, or refuse standard therapy
  * For those patients receiving phlebotomy only, the frequency over the past year must be at least one phlebotomy every 3 months.
* Undergone phlebotomy and attained a Hct < 47% (men) or < 45% (women) (or pre-specified Hct count that is tolerable) within 14 days prior to the start of study treatment
* Cessation of myelosuppressive agents prior to initiation of study treatment (unless approved by Geron Medical Monitor for unusual circumstances)

  * Hydroxyurea or anagrelide: Cessation 1 day prior to initiation of study treatment. Consideration to the timing of cessation of this therapy prior to the start of study treatment should take into account the requirement for phlebotomy.
  * INF-α or pegylated- INF-α: Cessation 4 weeks prior to initiation of study treatment
* Laboratory criteria (within 14 days of first study drug administration):

  * Platelets > the lower limit of normal (LLN)
  * ANC ≥ 1500/μL

General Criteria (All Patients)

* Willing and able to sign an informed consent
* Male or female, aged 18 years or older
* ECOG performance status 0-2
* Laboratory criteria (within 14 days of first study drug administration):

  * INR (or PT) and aPTT < 1.5 x the upper limit of normal (ULN)
  * Serum creatinine ≤ 2 mg/dL
  * Serum bilirubin < 2.0 mg/dL (patients with Gilbert's syndrome: serum bilirubin < 3 x ULN)
  * AST (SGOT) and ALT (SGPT) ≤ 2.5 x ULN
  * Alkaline phosphatase < 2.5 x ULN
* Any clinically significant toxicity from previous cancer treatments and/or major surgery must have recovered to Grade 0-1 prior to initiation of study treatment
* Women of childbearing potential must have a negative pregnancy test and agree to use effective birth control during and for at least 12 weeks after the last study treatment with imetelstat
* Male patients must agree to use effective birth control for themselves or their partner during and for 12 weeks after the last study treatment with imetelstat.

Exclusion Criteria

Patients who meet any of the following criteria will be excluded from screening and study entry:

* Women who are pregnant or breast feeding
* Prior stem cell transplantation
* Investigational therapy within 4 weeks prior to first study drug administration
* Clinically significant cardiovascular disease or condition including:

  * Uncontrolled congestive heart failure (CHF)
  * Need for anti-arrhythmic therapy for a ventricular arrhythmia
  * Clinically significant severe conduction disturbance per the Investigator's discretion
  * Ongoing angina pectoris requiring therapy
  * New York Heart Association (NYHA) Class II, III, or IV cardiovascular disease (see Appendix E)
* Known positive serology for human immunodeficiency virus (HIV)
* Serious co-morbid medical conditions, including active or chronically recurrent bleeding, clinically relevant active infection, cirrhosis, and chronic obstructive or chronic restrictive pulmonary disease per the Investigator's discretion
* Any other severe, acute, or chronic medical or psychiatric condition, laboratory abnormality, or difficulty complying with protocol requirements that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Investigator, would make the patient inappropriate for this study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2010-12; Primary Completion 2013-10 (Actual); Study Completion 2015-04 (Actual)

PRIMARY OUTCOMES:
Hematologic Response | From time of first dose (cycle 1 day 1) through end of study (12 mos after last participant is dosed)
  Primary objectives are as follows: ET patients - best hematologic response within the first year of therapy and PV patients - maintenance of Hct < 45% in men and < 42% in women (or pre-specified Hct count that is tolerable) without phlebotomy or myelosuppressive therapy within the first year of therapy. Secondary objectives, to determine the durability of hematologic response and to determine the rate of phlebotomy required within the first year of therapy.

SECONDARY OUTCOMES:
Safety and tolerability: Number of Patients with Hematological Toxicities, Non-Heme Grade 3 and 4 AEs, and Hemorrhagic Events | From time of first dose (cycle 1 day 1) through end of study (12 mos after last paricipant is dosed)
  The safety and tolerability of imtelstat will be assessed by the incidence, nature, relatedness and severity of adverse events, laboratory abnormalities and vital signs.

CONTACTS AND LOCATIONS:
Locations (12):
- United States (6):
  - City of Hope, Duarte, California
  - MDACC - Orlando, Orlando, Florida
  - University of Chicago, Chicago, Illinois
  - Johns Hopkins University - Bunting Blaustein Cancer Research Building, Baltimore, Maryland
  - Saint Francis Hospital, Greenville, South Carolina
  - MD Anderson Cancer Center, Houston, Texas
- Germany (5):
  - University Hospital of Essen - West German Cancer Center, Essen
  - Medizinische Klinik II, Abt. Hämatologie und Onkologie - Johann Wolfgang Goethe Universität, Frankfurt
  - SLK-Kliniken GmbH, Heilbronn
  - Hematology Oncology Center - Ludwig-Maximilians, University Munich Medical School, Munich
  - University Hospital Regensburg - Uniklinik Regensburg, Regensburg
- INSELSPITAL, University Hospital Bern, Bern, Switzerland

REFERENCES:
- [Derived] Oppliger Leibundgut E, Haubitz M, Burington B, Ottmann OG, Spitzer G, Odenike O, McDevitt MA, Roth A, Snyder DS, Baerlocher GM. Dynamics of mutations in patients with essential thrombocythemia treated with imetelstat. Haematologica. 2021 Sep 1;106(9):2397-2404. doi: 10.3324/haematol.2020.252817. PMID 32732354
- [Derived] Baerlocher GM, Oppliger Leibundgut E, Ottmann OG, Spitzer G, Odenike O, McDevitt MA, Roth A, Daskalakis M, Burington B, Stuart M, Snyder DS. Telomerase Inhibitor Imetelstat in Patients with Essential Thrombocythemia. N Engl J Med. 2015 Sep 3;373(10):920-8. doi: 10.1056/NEJMoa1503479. PMID 26332546